CLINICAL TRIAL: NCT01669408
Title: A Randomized Controlled Trial Evaluating Cold Infusions for Prehospital Induction of Cooling in Awake Stroke Patients (PreCOOL 1)
Brief Title: Prehospital COOLing 1 (PreCOOL 1)
Acronym: PreCOOL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. Sven Poli, Dr. Sven Poli, Consultant Neurologist, Principical Investigator, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PreCOOL 1
Record Dates: First submitted 2012-08-14; First posted 2012-08-21 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Stroke
Keywords: ischemic stroke; hemorrhagic stroke; prehospital cooling; induction of cooling; ambulance; emergency room; cold infusions; hypothermia; normothermia
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Emergencies; Hypothermia | interventions — Sodium Chloride; Ringer's Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cold infusions (Active Comparator): Infusion of 1L cold crystalloid solution (4°C) over 15 minutes
  Interventions: Drug: Cold crystalloid infusions, 0.9%NaCl or Ringer's solution
- Control group (No Intervention): Best medical treatment following international stroke guidelines

INTERVENTIONS:
Drug: Cold crystalloid infusions, 0.9%NaCl or Ringer's solution — Infusion of 1L cold crystalloid solution (4°C) over 15 minutes
  Arms: Cold infusions

SUMMARY:
Elevated body temperature was shown to be associated with worse outcome in acute stroke patients. PreCOOL 1 aims to investigate efficacy, feasibility and safety of prehospital cooling with cold infusions in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Suspected stroke
* Symptom onset ≤ 7 days
* Tympanic temperature ≥ 36.7°C
* Informed consent by the patient
* Age ≥ 18 years

Exclusion Criteria:

* Severe cardiac insufficiency (NYHA ≥ III)
* New anisocoria, severe nausea, vomiting or headache
* High-grade heart valve stenosis or insufficiency
* Acute pulmonary embolism
* Acute myocardial infarction
* Threatening ventricular dysrhythmia
* Known hematologic disease with increased risk of thrombosis (e.g. cryoglobulinemia, cold agglutinins, sickle cell anemia)
* Known vasospastic vascular disorder (e.g. Raynaud's phenomenon or thromboangiitis obliterans)
* Severe renal insufficiency with reduced diuresis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Tympanic Temperature | from randomization (prehospital) until arrival in the ER, an expected average of 45min
  Primary endpoint: Change of tympanic temperature between measurements before prehospital start of cooling an at arrival in the emergency room.

SECONDARY OUTCOMES:
Efficacy | single measurement at arrival in the ER
  Secondary efficacy endpoint: Proportion of patients having a oral temperature between 36 and 37.1°C at arrival in the ER.
Vital parameters | from randomization (prehospital) until arrival in the ER, an expected average of 45min
  Effects on vital parameters (e.g. HR, ECG, BP, SpO2) are registered.
Tolerability | from randomization (prehospital) until arrival in the ER, an expected average of 45min
  Tolerability outcome measures include the Bedside Shivering Assessment Scale (BSAS) and a 10 point visual analog scale to assess "feeling cold" and "shivering".
Safety | from randomization (prehospital) until first neuroimaging (ER), an expected average of 80min
  Safety outcome measures include the analysis of (severe) adverse events (e.g. bleeding complications, cardiac decompensation), dose of co-medication needed (e.g. antihypertensives, diuretics, anti-shivering medication), number of patients with oral temperature < 36°C and safety laboratory (Na, K, creatinine, urea, GFR, CK, CK-MB, troponin T, glucose, blood count, INR, aPTT, TT, NT-ProBNP and D-dimer)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Poli, Dr. med., Principal Investigator — University Hospital Heidelberg; Erik Popp, PD Dr. med., Principal Investigator — University Hospital Heidelberg
Locations (1):
- Rescue service, Dept. of Anesthesiology, University Hospital Heidelberg, Heidelberg, Germany